CLINICAL TRIAL: NCT07111728
Title: Multimodal Hyperspectral Imaging and Raman Spectroscopy for Intraoperative Assessment of Breast Tumor Resection Margins
Brief Title: Intraoperative Margin Assessment in Breast Cancer With HSI-Raman
Acronym: Spectra-BREAST
Status: Not yet recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Fabio Corsi, Prof., Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 0012251/25
Record Dates: First submitted 2025-07-28; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Breast-conserving surgery; Breast Cancer; Surgical margin assessment; Hyperspectral imaging; Raman spectroscopy; Optical spectroscopy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- DCIS breast cancer
  Interventions: Diagnostic Test: Spectra-BREAST system in DCIS Breast Cancer
- Invasive Breast Cancer
  Interventions: Diagnostic Test: Spectra-BREAST system in Invasive Breast Cancer

INTERVENTIONS:
Diagnostic Test: Spectra-BREAST system in Invasive Breast Cancer — Participants' excised breast lumpectomy specimens will be immediately imaged ex vivo using the investigational Spectra-BREAST system, a handheld optical device integrating two modalities
  Hyperspectral imaging (HSI):
  HSI captures reflectance spectra across 400-1400 nm over the entire specimen surface (up to 5 × 5 cm field of view). HIS provides spatial maps of tissue chemical composition and morphology to highlight regions suspicious for residual carcinoma.
  Point-wise Raman spectroscopy (RS):
  RS will allow to acquire high-resolution molecular fingerprints both at high and low Raman shift on selected "hotspots" flagged by HSI as at risk. RS will be acquired on the surface of the specimens confirming the possible presence of positive margins
  Spectra-BREAST system will allow to provide a near real time feedback to the surgeon on the presence and position of positive margins allowing a further resection if tissue if needed.
  Groups: Invasive Breast Cancer
Diagnostic Test: Spectra-BREAST system in DCIS Breast Cancer — Participants' excised breast lumpectomy specimens will be immediately imaged ex vivo using the investigational Spectra-BREAST system, a handheld optical device integrating two modalities Hyperspectral imaging (HSI): HSI captures reflectance spectra across 400-1400 nm over the entire specimen surface (up to 5 × 5 cm field of view). HIS provides spatial maps of tissue chemical composition and morphology to highlight regions suspicious for residual carcinoma. Point-wise Raman spectroscopy (RS): RS will allow to acquire high-resolution molecular fingerprints both at high and low Raman shift on selected "hotspots" flagged by HSI as at risk. RS will be acquired on the surface of the specimens and using a special needle probe 2 mm below the tissue surface thus confirming the possible presence of positive margins.
  Spectra-BREAST system will allow to provide a near real time feedback to the surgeon on the presence and position of positive margins allowing a further resection if tissue if needed
  Groups: DCIS breast cancer

SUMMARY:
Breast-conserving surgery (lumpectomy) aims to remove cancer while preserving healthy tissue, but up to 20% of patients require a second operation because cancer cells remain at the edge (margin) of the removed tissue. The Spectra-BREAST study evaluates a new optical device that combines hyperspectral imaging (HIS) and Raman spectroscopy (RS) with artificial-intelligence analysis to quickly assess the entire surface of excised breast specimens during surgery. By flagging areas at risk of positive margins in real time, the device may help surgeons remove any remaining cancer in a single procedure.

In this prospective, single-arm diagnostic study, surgeons will use the Spectra-BREAST system on freshly resected breast tissue from up to 99 women undergoing lumpectomy for invasive carcinoma or ductal carcinoma in situ. First, the device's cancer-detection algorithms will be trained on 74 specimens with known pathology. Then, in a separate group of patients, the fully integrated device will be tested on all six faces of each lumpectomy specimen and its predictions will be compared against the gold-standard histopathology margin assessment. Key measures include the sensitivity and specificity of the device's margin predictions, the time needed to generate results, and the device's usability in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of ductal carcinoma in situ (B5a) or invasive breast carcinoma (B5b) on pre-operative core needle biopsy

Scheduled to undergo breast-conserving surgery (lumpectomy)

Able and willing to provide written informed consent

Exclusion Criteria:

Pre-operative histologic or cytologic diagnosis of a benign breast lesion (B2/C2)

Initial diagnosis of advanced (stage III/IV) or metastatic breast carcinoma, or indication for neoadjuvant chemotherapy

Neurocognitive disorders that would impair comprehension of the study procedures or consent process

Concurrent pregnancy or breastfeeding

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All female patients referred consecutively to the Breast Unit at Istituti Clinici Scientifici Maugeri (IRCCS) in Pavia who present with an imaging-detected, clinically non-palpable breast lesion and are scheduled for breast-conserving surgery (lumpectomy).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of Spectra-BREAST system margin status prediction | Within 21 days after surgery (latest expected receipt of the final pathology report).
  Proportion of resection faces correctly classified by the Spectra-BREAST device as "positive margin" or "negative margin" when compared to gold-standard postoperative histopathology. Sensitivity and specificity will both be calculated independently in Invasive Breast Cancer and in DCIS breast cancer across all specimens in the validation cohort.

SECONDARY OUTCOMES:
Concordance of HSI-only versus combined HSI + RS predictions | During Spectra-BREAST procedure
  Percentage agreement between margin classifications made using hyperspectral imaging alone and those made by the integrated HSI + Raman spectroscopy algorithm, relative to histopathology results.
Time from specimen removal to Spectra-BREAST system result | Per specimen, measured intraoperatively
  Time (in minutes) from excision of the lumpectomy specimen to presentation of the Spectra-BREAST margin results.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo F Morasso, Ph.D., Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- Istituti Clinici Scientifici Maugeri IRCCS, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Official webpage of the Spectra-BREAST project — https://spectrabreast.eu/